CLINICAL TRIAL: NCT03283579
Title: Prenatal Omega-6/Omega-3 Ratio and Attention Deficit and Hyperactivity Disorder Symptoms in Children: a Population-based Longitudinal Study
Brief Title: Fatty Acids and Attention Deficit and Hyperactivity Disorder Symptoms
Status: Completed | Type: Observational
Sponsor: Barcelona Institute for Global Health (Other)
Responsible Party: Sponsor
Other Study IDs: mlopez
Record Dates: First submitted 2017-09-13; First posted 2017-09-14 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2017-09

CONDITIONS: Child Behavior Problem; Attention Deficit Hyperactivity Disorder; Fatty Acid Deficiency
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women

SUMMARY:
This study aimed to evaluate the longitudinal association between n-6:n-3 LCPUFAs ratio in cord blood and child ADHD symptoms at 4 and 7 years old. This study was based on the INMA project, a population-based birth cohort in Spain. Higher cord blood n-6:n-3 ratio was associated with higher subclinical ADHD symptoms during early and mid-childhood.

ELIGIBILITY:
Inclusion criteria:

* Age 16 years or older
* Singleton pregnancy
* No use of assisted reproductive techniques
* Intention to deliver at the reference hospital
* Ability to speak and understand Spanish or a local language

Ages: 4 Years to 8 Years | Sex: All
Age Groups: Child
Study Population: This study was based on data from a population-based birth cohort, INMA (Infancia y Medio Ambiente [Environment and Childhood]) project, including four Spanish regions: Asturias (n=494) and Gipuzkoa (Basque Country) (n=638) on the Cantabrian coast, and Sabadell (Catalonia) (n=657) and Valencia (n=855) on the Mediterranean coast.
Sampling Method: Non-Probability Sample
Enrollment: 2644 (Actual)
Dates: Start 2003-11 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Fatty acid ratio in cord blood | 2004-2008
ADHD 4 years old | 2008-2012
ADHD 7 years old | 2012-2016

IPD SHARING:
Plan to Share IPD: No